CLINICAL TRIAL: NCT00343889
Title: Immunogenicity Study of a DTaP-Hep B-PRP-T Combined Vaccine Compared to Tritanrix-HepB/Hib™, Both Given Concomitantly With the Oral Polio Vaccine at 6, 10, and 14 Weeks of Age in Healthy Infants in the Philippines
Brief Title: Comparison of DTaP-HB-PRP~T Combined Vaccine to Tritanrix-HepB/Hib™, Both Given Concomitantly With Oral Polio Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AL203
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Infections
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B Hansenula (HB); Haemophilus influenzae type b; Haemophilus Influenzae
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-Hib-hepatitis B vaccine; Poliovirus Vaccine, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: DTaP-Hep B-PRP-T + Oral Polio Vaccine (OPV) vaccine (Experimental): Participants received 3 doses of the DTaP-Hep B-PRP~T concomitantly with Oral Polio Vaccine (OPV), 1 dose each at 6, 10, and 14 weeks of age.
  Interventions: Biological: DTaP-HB-PRP~T vaccine + OPV; Biological: Oral Polio Vaccine
- Group 2: Tritanrix-HepB/Hib™ + OPV vaccine (Active Comparator): Participants received 3 doses of Tritanrix-Hep B/Hib™ concomitantly with Oral Polio Vaccine (OPV) at 6, 10, and 14 weeks of age.
  Interventions: Biological: Tritanrix-HepB/Hib™ + OPV vaccine; Biological: Oral Polio Vaccine

INTERVENTIONS:
Biological: DTaP-HB-PRP~T vaccine + OPV — 0.5 mL, Intramuscular
  Arms: Group 1: DTaP-Hep B-PRP-T + Oral Polio Vaccine (OPV) vaccine
Biological: Tritanrix-HepB/Hib™ + OPV vaccine — 0.5 mL, Intramuscular
  Arms: Group 2: Tritanrix-HepB/Hib™ + OPV vaccine
Biological: Oral Polio Vaccine — Oral co-administered with study vaccine

SUMMARY:
The purpose of this study is to support the registration of the pentavalent DTaP-HB-PRP~T vaccine in countries that follow the World Health Organization-Expanded Program of Immunization (WHO-EPI) schedule.

The primary objective is:

* To demonstrate that the pentavalent DTaP-HB-PRP~T combined vaccine does not induce a lower immune response than Tritanrix-HepB/Hib™ in terms of the seroprotection rate to hepatitis B (HB) one month after a 3-dose primary series at 6, 10, and 14 weeks of age.

The secondary objectives are:

* To describe in each group the immunogenicity parameters one month after the 3-dose primary series at 6, 10, and 14 weeks of age; and
* To evaluate the overall safety in terms of any adverse events in the first 28 days after each injection and any serious adverse events during the entire trial.

ELIGIBILITY:
Inclusion Criteria:

* Six week old infants (42 to 50 days old) on the day of inclusion; of either gender.
* Mother tested as seronegative for hepatitis B surface antigen (HBsAg) between 28 weeks of pregnancy and up to 4 days after delivery
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by one parent or other legal representative if appropriate (independent witness is mandatory if parent is illiterate)
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency; immunosuppressive therapy such as long-term systemic corticosteroid therapy.
* Chronic illness at a stage that could interfere with the conduct or completion of the trial
* Blood or blood-derived products received since birth
* HB vaccination since birth
* Any vaccination in the four weeks preceding the first trial vaccination
* Any planned vaccination (except trial vaccines and bacillus Calmette-Guerin (BCG) during the trial
* Documented history of pertussis, tetanus (T), diphtheria (D), polio, or Haemophilus influenzae type b (Hib) infection(s) (confirmed either clinically, serologically, or microbiologically)
* Known personal or maternal history of HIV, HBsAg or hepatitis C seropositivity
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular (IM) vaccination
* History of seizures
* Febrile (rectal temperature ≥ 38.0°C) or acute illness on the day of inclusion.

Ages: 42 Days to 50 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 379 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Philippines (2):
  - Manila
  - Quezon City

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 07 July 2006 to 26 September 2006 in 2 clinical centers in the Philippines.
Pre-assignment Details: A total of 379 participants who met all the inclusion and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received 3 doses of the DTaP-Hep B-PRP~T concomitantly with Oral Polio Vaccine (OPV), 1 dose each at 6, 10, and 14 weeks of age.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received 3 doses of Tritanrix-Hep B/ Hib™ concomitantly with Oral Polio Vaccine (OPV) at 6, 10 and 14 weeks of age.
Period: Overall Study
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Started | 190 | 189
Completed | 187 | 188
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV | Total
Number analyzed (Participants) | 190 | 189 | 379
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 190 | 189 | 379
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Weeks] | 6.31 (0.308) | 6.31 (0.304) | 6.31 (0.306)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 92 | 193
  Male | 89 | 97 | 186
Region of Enrollment [Number; unit: Participants]
  Philippines | 190 | 189 | 379

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Anti-Hepatitis B Responses After Vaccination With Either DTaP-Hep B-PRP~T Concomitantly With Oral Polio Vaccine (OPV) or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for hepatitis B (HBs) antibodies.
  Anti-Hepatitis B Responses was defined as titers ≥ 100 mIU/mL at 30 days after the third vaccination.
Time Frame: 1 month post third vaccination
Population: Anti-Hepatitis B Responses was assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 184 | 186
Participants | 54 | 97

2. Primary Outcome: Number of Participants With Seroprotection to Hepatitis H Antigen After Vaccination With Either DTaP-Hep B-PRP~T Concomitantly With Oral Polio Vaccine (OPV) or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for hepatitis B (HBs) antibodies.
  Seroprotection was defined as titers ≥ 10 mIU/mL at 30 days after the third vaccination.
Time Frame: 1 month post third vaccination
Population: Seroprotection to hepatitis H Antigen was assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 184 | 186
Participants | 146 | 167

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies After Vaccination With Either DTaP-Hep B-PRP-T Concomitantly With OPV or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity were assessed by means of enzyme immunoassay (EIA) for antibodies to the vaccine antigens 1 month after the third vaccination (Day 150).
Time Frame: 1 month post third vaccination
Population: Geometric Mean Titers (GMTs) of Vaccine Antibodies were assessed in the per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 260 | 271
Titers
  Anti-Hepatitis B (N = 184, 186) | 39.1 [31.0 to 49.2] | 86.2 [68.0 to 109]
  Anti-PRP (N = 178, 185) | 2.35 [1.83 to 3.01] | 7.82 [6.45 to 9.48]
  Anti-Diphtheria (N = 184, 186) | 0.018 [0.015 to 0.022] | 0.018 [0.014 to 0.021]
  Anti-Tetanus (N = 184, 186) | 1.30 [1.16 to 1.46] | 1.76 [1.58 to 1.97]
  Anti-Pertussis (N = 183, 184) | 5.16 [4.36 to 6.11] | 5.84 [4.81 to 7.09]
  Anti-Filamentous Hemagglutinin (N = 184, 186) | 5.50 [4.68 to 6.48] | 5.71 [4.85 to 6.71]

4. Secondary Outcome: Number of Participants With Anti-Diphtheria and Anti-Tetanus Responses After Vaccination With Either DTaP-Hep B-PRP~T Concomitantly With Oral Polio Vaccine (OPV) or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for Diphtheria and Tetanus antibodies.
  Anti-Diphtheria and anti-tetanus Responses were assayed at ≥ 0.01 IU/mL and at ≥ 0.1 IU/mL at 30 days after the third vaccination.
Time Frame: 1 month post third vaccination
Population: Anti-Hepatitis B Responses was assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 184 | 186
Participants
  Anti-Diphtheria ≥ 0.01 IU/mL | 137 | 134
  Anti-Diphtheria ≥ 0.1 IU/mL | 13 | 11
  Anti-Tetanus ≥ 0.01 IU/mL | 184 | 186
  Anti-Tetanus ≥ 0.1 IU/mL | 184 | 186

5. Secondary Outcome: Number of Participants With Seroconversion for Anti-Pertussis and Anti-Filamentous Hemagglutinin Antibodies After Vaccination With Either DTaP-Hep B-PRP-T Concomitantly With OPV or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Anti-Pertussis toxoid and Anti-Filamentous Hemagglutinin antibodies were assessed by means of enzyme immunoassay (EIA).
  Seroconversion was defined as ≥ 4 fold increase in antibody titers from Day 0 to 30 days after the third vaccination.
Time Frame: 1 month post third vaccination
Population: Seroconversion for anti-Pertussis toxoid and anti-Filamentous Hemagglutinin antibodies were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 184 | 186
Participants
  Anti-Pertussis Toxoid (N =184, 180) | 183 | 168 [0 to 0]
  Anti-Filamentous Hemagglutinin (N = 178, 131) | 178 | 116 [0 to 0]

6. Secondary Outcome: Number of Participants Reporting At Least One Solicited Injection Site and Systemic Reaction Following Each Vaccination With Either DTaP-Hep B-PRP-T Concomitantly With Oral Polio Vaccine (OPV) or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling; Systemic reactions: Fever (Temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability.
  Grade 3 reactions defined as: Tenderness - cries when injected limb is moved; Erythema and Swelling - ≥ 5cm; Fever - temperature ≥ 39.6ºC; Vomiting - ≥6 episodes per 24 hours; Crying - inconsolable crying for >3 hours; Somnolence - sleeping most of the time or difficulty to wake up; Anorexia - refuses ≥3 feeds; and Irritability - inconsolable.
Time Frame: Day 0 up to Day 7 after each vaccination
Population: Safety was assessed on the safety analysis (intent-to-treat) population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 190 | 189
Participants
  Injection site Pain post any vaccination | 123 | 152 [0 to 0]
  Grade 3 Injection site Pain post any vaccination | 7 | 24 [0 to 0]
  Injection site Pain post-vaccination 1 | 100 | 142 [0 to 0]
  Injection site Pain post-vaccination 2 | 86 | 109 [0 to 0]
  Injection site Pain post-vaccination 3 | 62 | 88 [0 to 0]
  Injection site Erythema post any vaccination | 121 | 148 [0 to 0]
  Grade 3 Injec. site Erythema post any vaccination | 2 | 3 [0 to 0]
  Injection site Erythema post-vaccination 1 | 70 | 89 [0 to 0]
  Injection site Erythema post-vaccination 2 | 70 | 105 [0 to 0]
  Injection site Erythema post-vaccination 3 | 76 | 104 [0 to 0]
  Injection site Swelling post any vaccination | 60 | 107 [0 to 0]
  Grade 3 Injec. site Swelling post any vaccination | 4 | 7 [0 to 0]
  Injection site Swelling post-vaccination 1 | 41 | 89 [0 to 0]
  Injection site Swelling post-vaccination 2 | 28 | 57 [0 to 0]
  Injection site Swelling post-vaccination 3 | 24 | 49 [0 to 0]
  Pyrexia post any vaccination | 85 | 129 [0 to 0]
  Grade 3 Pyrexia post any vaccination | 1 | 4 [0 to 0]
  Pyrexia post-vaccination 1 | 59 | 106 [0 to 0]
  Pyrexia post-vaccination 2 | 40 | 54 [0 to 0]
  Pyrexia post-vaccination 3 | 22 | 51 [0 to 0]
  Vomiting post any vaccination | 43 | 61 [0 to 0]
  Grade 3 Vomiting post any vaccination | 0 | 0 [0 to 0]
  Vomiting post-vaccination 1 | 37 | 40 [0 to 0]
  Vomiting post-vaccination 2 | 16 | 24 [0 to 0]
  Vomiting post-vaccination 3 | 9 | 13
  Crying post any vaccination | 56 | 97
  Grade 3 Crying post any vaccination | 0 | 0
  Crying post-vaccination 1 | 41 | 71
  Crying post-vaccination 2 | 29 | 42
  Crying post-vaccination 3 | 16 | 34
  Somnolence post any vaccination | 52 | 63
  Grade 3 Somnolence post any vaccination | 2 | 2
  Somnolence post-vaccination 1 | 43 | 49
  Somnolence post-vaccination 2 | 24 | 26
  Somnolence post-vaccination 3 | 10 | 18
  Anorexia post any vaccination | 48 | 67
  Grade 3 Anorexia post any vaccination | 1 | 1
  Anorexia post-vaccination 1 | 32 | 50
  Anorexia post-vaccination 2 | 20 | 25
  Anorexia post-vaccination 3 | 16 | 27
  Irritability post any vaccination | 102 | 128
  Grade 3 Irritability post any vaccination | 4 | 7
  Irritability post-vaccination 1 | 90 | 116
  Irritability post-vaccination 2 | 48 | 71
  Irritability post-vaccination 3 | 32 | 56

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 238 post-vaccination.
Description: The total number (N) for each adverse event indicated those with available data for the event.
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Serious Adverse Events (participants affected / at risk) | 17/190 | 10/189
Other Adverse Events (participants affected / at risk) | 123/190 | 152/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=190) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=189)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bullus impetigo (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (8) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=190) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=189)
Vomiting (Gastrointestinal disorders) | 43/189 | 61
Injection site pain (Gastrointestinal disorders) | 123/189 | 152
Injection site erythemia (General disorders) | 121/189 | 148
Injection site swelling (General disorders) | 60/189 | 107
Pyrexia (General disorders) | 85/189 | 129
Pyrexia (General disorders) | 7 | 17
Anorexia (Metabolism and nutrition disorders) | 48/189 | 67
Somnolence (Nervous system disorders) | 52/189 | 63
Upper respiratory tract infection (Infections and infestations) | 89 | 113
Rhinitis (Metabolism and nutrition disorders) | 14 | 16
Crying (Psychiatric disorders) | 56/189 | 97
Irritability (Psychiatric disorders) | 102/189 | 128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications